CLINICAL TRIAL: NCT01001325
Title: A Randomized Controlled Trial of the Effect of Seasonal Influenza Vaccination on the Incidence of Infection Due to the 2009 H1N1 Influenza
Brief Title: Does Seasonal Influenza Vaccination Affect the Incidence of pH1N1 Influenza?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: CRT113936
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Influenza
Keywords: influenza; vaccine; observer blind
MeSH Terms: conditions — Influenza, Human | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seasonal influenza vaccination (Experimental): Receipt of Fluviral seasonal (2009-2010, Canadian) influenza vaccination as per manufacturers specification
  Interventions: Biological: Fluviral influenza vaccine, 2009-2010
- Placebo (Placebo Comparator): 0.5 mL normal saline
  Interventions: Biological: Normal saline

INTERVENTIONS:
Biological: Fluviral influenza vaccine, 2009-2010 — 0.5 mL intramuscular
  Arms: Seasonal influenza vaccination
Biological: Normal saline — 0.5 mL intramuscular
  Arms: Placebo

SUMMARY:
Since the onset of the 2009 pandemic, several observational public health investigations in Canada have identified evidence that suggests that adults, particularly younger adults, who have previously received seasonal influenza vaccine are at increased risk of infection with the 2009 pandemic strain of H1N1 (pH1N1). Investigations in Australia, the United States and the United Kingdom have not identified this effect. While it is not possible to have an answer to whether this affect is real prior to the second wave of the 2009 pandemic, it remains vital to future influenza vaccination programs that the hypothesis that, in 2009, seasonal vaccine increases or decreases the risk of pH1N1 infection be confirmed or refuted.

The objective of this study is to determine whether Ontario adults aged 18-60 years who receive the 2009 seasonal influenza vaccine will be at a 2 fold or greater increased risk of infection with influenza pH1N1 during the second or third wave of the 2009 pandemic.

DETAILED DESCRIPTION:
This study will be an observer -blind randomized controlled trial.

This study will primarily recruit patients from an existing cohort of adult health care and other workers in Toronto, as of September 15, 2009, almost 1000 adults are participating in this cohort; with approximately 75 new cohort members being recruited weekly (target is 1300). Recruitment will be supplemented by enrollment at Hamilton Health Sciences Centre (N~3920 employees plus physicians & midwives) and Queen Elizabeth II Health Centre in Halifax (N~6000 employees plus physicians & midwives).

To date, health care workers in the Toronto cohort have been recruited at the Mount Sinai Hospital, Toronto East General Hospital, and North York General Hospital. Recruitment is just beginning at Sunnybrook Health Sciences Centre, and the University Health Network.

Non-health care workers are being recruited from several large Toronto employers of primarily office workers. These include the Ontario Agency for Health Protection and Promotion, the head offices of the Ontario Power Generation Corporation, the Art Gallery of Ontario, and the head offices of Scotia Bank. Non-health care workers should meet inclusion criteria and should not work primarily with children or from a home office.

Participants in the study are completing web-based diaries weekly, and, whenever they develop symptoms possibly compatible with influenza, are submitting nasal swabs, and completing symptom diaries daily while ill. Nasal swabs are tested by polymerase chain reaction (PCR) on a same or next day basis with antivirals prescribed to participants who develop influenza.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 60 years old, inclusive, as of September 1st, 2009;
2. understand the study, agree to its provisions, and give written informed consent prior to entry;
3. available for follow-up during the study period;
4. have convenient access to a computer with internet access and basic skills for use of the internet;

Exclusion Criteria:

1. planning to spend more than two consecutive weeks outside of Canada from October 1, 2009 to April 15th 2010.
2. received immunoglobulin within six months of study entry;
3. has already received a 2009 seasonal influenza vaccine (southern or northern hemisphere)
4. has had laboratory-confirmed infection with 2009 H1N1 influenza
5. is participating in a clinical trial that would result in the receipt of investigational medication during the study period;
6. allergic to eggs, to influenza vaccine, or any components of the seasonal influenza vaccine
7. has had a previous severe adverse event associated with an influenza vaccine
8. has a significant chronic underlying illness that would warrant seasonal influenza vaccine in a usual year, or is known to be pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 468 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison J McGeer, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Brenda L. Coleman, PhD, Principal Investigator — MOUNT SINAI HOSPITAL; Natasha Crowcroft, MD, Principal Investigator — Ontario Agency for Health Protection & Promotion; Karen Green, MSc, Study Director — MOUNT SINAI HOSPITAL; Kevin Katz, MD, Study Director — North York General Hospital; Mark Loeb, MD, Study Director — Hamilton Health Sciences Centre; Donald Low, MD, Study Director — MOUNT SINAI HOSPITAL; Shelly McNeil, MD, Study Director — Queen Elizabeth II Health Sciences Centre; Matthew Muller, MD, PhD, Study Director — Unity Health Toronto; Andrew Simor, MD, Study Director — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - North York General Hospital, North York, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolment start: October 5, 2009 Enrolment complete: February 3, 2010
  Enrolment was conducted from a variety of work places and university settings.
Period: Overall Study
Arm/Group | Seasonal Influenza Vaccination | Placebo
Started | 234 | 234
Completed | 216 | 224
Not Completed | 18 | 10
Not completed — Lost to Follow-up | 16 | 10
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seasonal Influenza Vaccination | Placebo | Total
Number analyzed (Participants) | 234 | 234 | 468
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 233 | 234 | 467
  >=65 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 36.8 (12.6) | 35.7 (12.5) | 36.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 157 | 305
  Male | 86 | 77 | 163
Region of Enrollment [Number; unit: participants]
  Canada | 234 | 234 | 468

OUTCOME MEASURES:

1. Primary Outcome: Number of pH1N1 Influenza Infections as Diagnosed by PCR From Mid-turbinate Swab
Description: Influenza infection (pH1N1) as diagnosed by PCR from self-collected mid-turbinate swab. Participant is asked to collect a swab when they have symptoms possibly compatible with an acute viral respiratory illness: 1) fever without another obvious source, 2) at least two new respiratory symptoms (runny or stuffy nose, sneezing, sore or scratchy throat, hoarseness, cough), or 3) one respiratory symptom (as above) and one systemic symptom (fever, malaise, muscle aches, headache, fatigue)
Time Frame: day +7 post seasonal influenza vaccination (or placebo) to end of study
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Seasonal Influenza Vaccination | Placebo
Number analyzed (Participants) | 234 | 234
participants | 2 [0.23 to 6.55] | 4 [1.17 to 9.59]
Statistical Analysis 1: Comparison: Seasonal Influenza Vaccination vs Placebo; Null hypothesis: There is no difference in incidence of pandemic strain influenza infection for people given seasonal influenza vaccine compared to those given a placebo. Power to detect a 2-fold difference if attack rate in non-vaccinated participants is 10%: 86%; Test type: Superiority or Other; p = 0.685, Fisher Exact

ADVERSE EVENTS:
Time Frame: Enrolment to March 28, 2010 - Maximum: 6 months
Arm/Group | Seasonal Influenza Vaccination | Placebo
Serious Adverse Events (participants affected / at risk) | 1/234 | 1/234
Other Adverse Events (participants affected / at risk) | 0/234 | 0/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seasonal Influenza Vaccination (N=234) | Placebo (N=234)
death (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — Not related to study drug
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
A major limitation to this study was the date of enrolment for the subjects: only 249 (53%) of the subjects were enrolled by the end of second wave of the pandemic (and a third wave did not occur before the end of the study).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less